CLINICAL TRIAL: NCT06363721
Title: A Pilot Study of a Commercially-available Oil Rinse Product (PerioPull™) on Markers of Dental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Designs for Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DFH00125
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Oral Health

STUDY DESIGN:
Intervention Model Description: The proposed study is a 12-week pilot study of PerioPull™. Eligible participants will be recruited from within the clinical practice of the periodontist. All study outcomes will be measurements and testing during three dental visits spaced 6 weeks apart. These are typical assessments in routine clinical practice. All study outcomes are described in detail in an ensuing section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PerioPull™ (Experimental): Participants will swish 1 teaspoon (approx. 5 mL) of oil in the mouth for a minimum of 5 minutes after their normal brushing routine, as is suggested on the label of the bottle. They will spit out the oil and not rinse to allow for longer contact to the teeth and gums. This will be once a day for 12 weeks.
  Interventions: Dietary Supplement: PerioPull™

INTERVENTIONS:
Dietary Supplement: PerioPull™ — PerioPull™ is a natural oil rinse formula to support overall oral/gum health, tooth stains, and natural teeth whitening. PerioPull™ includes Medium Chain Triglycerides (C8, C10, C12) (from coconut oil), Bixa orellana (Annatto) Seed Extract (GG-Gold®), Natural Mint Flavor, Bromelain, Ubiquinone, Delta Tocotrienols.

SUMMARY:
The primary purpose of this study is to evaluate the impact of a commercially-available oil rinse product (PerioPull™) on parameters of dental health among a sample of adults. PerioPull™ is commercially available and sold primarily from clinicians' offices.

A 12-week pilot study will be conducted to achieve the purpose of this study. The research team hypothesizes that PerioPull™ will improve a variety of validated markers of dental health that are commonly used in clinical practice.

DETAILED DESCRIPTION:
Patients that suffer from dental health issues often have a deeper than normal pocket depth. These pockets can become filled with infection causing bacteria causing inflammation around the tooth leading to periodontal disease.

The current recommendations are to brush with Sensodyne, use a special mouthwash, do not brush as hard, or use an electric toothbrush.

PerioPull™ is a natural oil rinse formula to support overall oral/gum health, tooth stains, and natural teeth whitening. This formula contains specific nutrients that have been previously studied and shown to be efficacious in oral health These actions do not have any known side effects, which present an advantage over standard dental treatments with fluoride, chlorhexidine, hydrogen peroxide and other chemicals.

This oil rinse formula is a commercially available product sold primarily from physicians' offices. As indicated in the ingredient list provided below, PerioPull™ includes Medium Chain Triglycerides (C8, C10, C12) (from coconut oil), Bixa orellana (Annatto) Seed Extract (GG-Gold®), Natural Mint Flavor, Bromelain, Ubiquionone, Delta Tocotrienols.

The proposed study is a 12-week pilot study of PerioPull™. Eligible participants will be recruited from within the clinical practice of the periodontist.

Study outcomes will consist of parameters of dental health among a sample of adults. These outcomes will be collected during a dental visit and assessed at baseline, six weeks, and at the conclusion of the 12-week clinical trial.

Oral samples that are obtained during clinical visits will be sent to lab utilized by participating clinical practices for analysis of study outcomes.

The outcomes in this clinical trial have been studied in previous clinical trials among dental patients. One oral sample at each of the three study visits is all that is required to collect outcomes.

All study outcomes will be measurements and testing during three dental visits spaced 6 weeks apart. These are typical assessments in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Plaque index of at least 1
* Gingival index of at least 1
* Pocket depth no greater than 5 mm
* Able to understand and write English
* Voluntarily consent to the study and understand its nature and purpose including potential risks and side effects
* Maintain current dental hygiene routine
* Bleeding on probing

Exclusion Criteria:

* Current daily use of any products containing the nutrients and/or herbs in the study product
* Known allergies to any substance in the study product
* Current daily tobacco smoker
* Currently pregnant or lactating women or women planning to become pregnant in the next 12 weeks
* Active oral infection (ie. herpes, candida)
* Recently on antibiotics (past 3 months)
* Undergone recent periodontal therapy (last 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Plaque Index | Baseline, 6 weeks, and 12 weeks
  Assesses the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth, except the third molars. The bacterial plaque developer solution was used to define cumulative amounts of plaque with criteria from 0 to 5. Once the values of the individual teeth are recorded, they are added and divided by the number of teeth examined to obtain the plaque index of each patient.
Gingival Index | Baseline, 6 weeks, and 12 weeks
  A method of recording the clinical severity of gingival inflammation. It is based upon probe measurement of periodontal pockets and on gingival tissue status.
Pocket Depth | Baseline, 6 weeks, and 12 weeks
  A measurement in millimeters of the depth from the gingival margin to the epithelial attachment in unhealthy gingival tissue. The pocket depth usually consists of depths great than 3 mm. pocket.

SECONDARY OUTCOMES:
Intraoral Photos | Baseline, 6 weeks, and 12 weeks
  Photos taken of the teeth, gums, and oral tissue. These may be a single tooth, a group of teeth, or any area of the mouth. Intraoral photos help establish a baseline for all dental conditions and are used as a tool to monitor any recession or suspicious lesions.
MyPerioPath® | Baseline, 6 weeks, and 12 weeks
  Used test for the detection of oral pathogens that cause gum disease and threaten oral & systemic health. It provides early warning of oral pathogens to enable the personalization of periodontal treatment. This test is non-invasive oral rinse collection (OralDNA® Labs)

CONTACTS AND LOCATIONS:
Locations (1):
- Julian Center for Comprehensive Dentistry, Ellicott City, Maryland, United States

IPD SHARING:
Plan to Share IPD: No